CLINICAL TRIAL: NCT01856075
Title: Relative Effectiveness of Dronedarone vs. Other Treatments of Atrial Fibrillation
Brief Title: Effectiveness Study of Atrial Fibrillation
Acronym: EFFECT-AF
Status: Completed | Type: Observational
Sponsor: La-ser Europe Limited (Other)
Responsible Party: Sponsor
Other Study IDs: Sanofi-EFFECT-AF
Record Dates: First submitted 2013-05-09; First posted 2013-05-17 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Dronedarone; Cohort; Effectiveness
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients treated with dronedarone: Patients treated with dronedarone at inclusion
- Patients treated with other antiarrhythmic drugs of interest: The antiarrhythmic drugs of interest to which dronedarone will be compared are:
  * Class 1a/1c antiarrhythmics
  * Sotalol
  * Amiodarone

SUMMARY:
This is an international observational multicentre study to be conducted in Germany, Spain, Italy and USA. The main objective of the study is to evaluate the relative effectiveness of dronedarone in real world clinical practice versus other anti-arrhythmic agents of interest. The design of the study is a historic-prospective cohort with dynamic exposure and stratified competitive recruitment with balanced comparison groups of dronedarone versus alternative antiarrhythmic drugs of interest.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years old or above
* Patient with paroxysmal or persistent atrial fibrillation
* Patient using an AAi (antiarrhythmic drug of interest) or dronedarone (index drug)
* Patient's treatment changed from one AAi to another AAi or dronedarone OR from no antiarrhythmic therapy to the start of AAi or dronedarone therapy during previous 6 months before the date of recruitment
* Patient with at least 6 months of medical and treatment information prior to the start of the index drug
* Patient able to answer the telephone interview in a language of the participating country: English, German, Italian or Spanish (with or without proxy).

Exclusion Criteria:

* Patient with heart failure (NYHA class IV)
* Patient with permanent Atrial Fibrillation
* Patient with psychiatric conditions preventing the participation to the study according to the physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an international observational multicentre study to be conducted in the following four countries: Germany, Spain, Italy and USA. Patients will be will be recruited from cardiology clinics, both hospital and non-hospital based, depending on particulars of treatment pathway of ppAF patients in each country.
Sampling Method: Non-Probability Sample
Enrollment: 1015 (Actual)
Dates: Start 2012-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline Recurrence of Atrial Fibrillation | 3 month; 6 month; 12-18 month
  Assessment of the recurrence of atrial fibrillation (change from baseline) at 3 month, 6 month, and 12-18 month of follow-up

SECONDARY OUTCOMES:
Change from baseline Cardiovascular hospitalisation | 3 month; 6 month; 12-18 month
Change from baseline AV node ablation and catheter ablation for Atrial Fibrillation | 3 month; 6 month; 12-18 month
Change from baseline Progression to permanent Atrial Fibrillation | 3 month; 6 month; 12-18 month
Change from baseline Clinical progression to heart failure and left ventricular systolic dysfunction | 3 month; 6 month; 12-18 month
Change from baseline Congestive heart failure | 3 month; 6 month; 12-18 month
Change from baseline Interstitial pulmonary disease | 3 month; 6 month; 12-18 month
Change from baseline Liver injury/toxicity | 3 month; 6 month; 12-18 month
Change from baseline Renal insufficiency/failure | 3 month; 6 month; 12-18 month
Change from baseline Cerebrovascular accident/Stroke | 3 month; 6 month; 12-18 month
Change from baseline Myocardial infarction | 3 month; 6 month; 12-18 month
Change from baseline Torsade de pointes | 3 month; 6 month; 12-18 month
Death | 3 month; 6 month; 12-18 month
  Assessed at each follow-up: 3 month, 6 month, and 12-18 month

CONTACTS AND LOCATIONS:
Overall Officials: Artak Khachatryan, PhD, Study Director — LA-SER Europe
Locations (1):
- Praxis fuer Kardiologie, Im Muehlenbach 2B, Bonn, Germany